CLINICAL TRIAL: NCT03625791
Title: Validation of a Genetic Signature to Predict the Development of Sarcomas
Acronym: PREDISARC
Status: Completed | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: PREDISARC
Record Dates: First submitted 2018-08-08; First posted 2018-08-10 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Genetic Signature in Development of Sarcomas
Keywords: sarcoma; genetic
MeSH Terms: conditions — Sarcoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- radiation-induced sarcomas
  Interventions: Biological: blood sample
- radiotherapy for at least 5 years and without sarcomas
  Interventions: Biological: blood sample
- primary sarcomas
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — 1 tube with 4 ml of blood per patient

SUMMARY:
The aim of the SARI study was to describe biomarkers of predisposition to the development of sarcomas in irradiated territory. This study included 120 patients with sarcoma in irradiated territory and 240 patients who had been treated with radiotherapy for more than 5 years and had not developed sarcoma.

Following the sequencing of the exomes of all these patients, the SARI study made it possible to highlight a genetic signature from 11 genes, predictive of the appearance of a sarcoma after a first radiotherapy. This signature is the subject of a patent (BFF 170286 / VF, filed on June 22, 2017). A final validation step with samples that have not been used to optimize this signature is now required. Moreover, it is now necessary to validate if this signature is specific to the predisposition to the development of radiation-induced sarcomas only or if this signature is also valid for the predisposition to the development of all sarcomas, even primary ones.

The objective of the PREDISARC study is to evaluate the specificity of this genetic signature (11 genes) with the appearance of sarcomas in irradiated territory compared to a population without sarcoma that has been treated with radiotherapy.

DETAILED DESCRIPTION:
A total of 60 patients will be included in this pilot study:

* Group 1: 20 patients with induced radio sarcoma
* Group 2: 20 patients without primary sarcoma or induced radio sarcoma
* Group 3: 20 patients with primary sarcoma These numbers will make it possible to have preliminary data making it possible to judge the interest of the genetic signature in the prediction of the radiation-induced sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient at the time of initial radiotherapy or diagnosis of primary sarcoma.
2. Patient belonging to one of these 3 groups :

   Group 1: Patient treated with radiotherapy for cancer other than primary sarcoma and who developed sarcoma (other than osteosarcoma) in the irradiated area.

   OR Group 2: Patient who received radiotherapy for more than 5 years and did not develop sarcoma or other secondary cancers OR Group 3: Patient who developed primary sarcoma and who had never been treated with radiotherapy
3. Patient who have signed informed consent to participate in the study.
4. Affiliation to the social security system.

Exclusion Criteria:

1. Patient unable to understand, read and / or sign informed consent.
2. Person benefiting from a protection system for adults (including guardianship and trusteeship)
3. Pregnant or lactating woman.
4. Patient who participated in the SARI study "Predictive study of sarcomas developed in irradiated territory from the GSF-GETO database (ID-RCB no .: 2011-A01102-39)"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Group 1: 20 patients with sarcoma developed in irradiated territory
  * Group 2: 20 patients treated for cancer by radiotherapy for more than 5 years and who have not developed sarcoma
  * Group 3: 20 patients with primary sarcoma
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2022-06-19 (Actual); Study Completion 2022-06-19 (Actual)

PRIMARY OUTCOMES:
DNA | at the inclusion
  Bioinformatic analyzes will be realized out blindly on the 11 genes of the signature to validate determining the group of belonging of the patients

CONTACTS AND LOCATIONS:
Overall Officials: Gilles TRUC, Principal Investigator — CGFL, Dijon
Locations (3):
- France (3):
  - Institu Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Institut Gustave Roussy, Villejuif